CLINICAL TRIAL: NCT02864498
Title: A Randomised, Double-blind, Placebo-controlled, Phase 2b Study to Assess the Efficacy and Safety of Orally Administered DS107 in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Efficacy and Safety Study of Orally Administered DS107 in Moderate to Severe Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DS Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS107G-03
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Results first posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-09

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1g DS107 (Experimental): 1g DS107 (2 DS107 capsules and 2 placebo capsules) orally administered once-daily for 8 weeks.
  Interventions: Drug: DS107
- 2g DS107 (Experimental): 2g DS107 (4 DS107 capsules) orally administered once-daily for 8 weeks.
  Interventions: Drug: DS107
- Placebo (Placebo Comparator): Placebo (4 placebo capsules) orally administered once-daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS107
  Arms: 1g DS107; 2g DS107
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether orally administered DS107 (1g and 2g doses) is effective in the treatment of moderate to severe atopic dermatitis.

Oral DS107 capsules will be administered for 8 weeks and will be compared against placebo.

The study will enroll approximately 300 subjects.

DETAILED DESCRIPTION:
The study will consist of 3 treatment arms, each consisting of approximately 100 subjects.

Treatment Arm 1 will receive 1g Oral DS107 daily. Treatment Arm 2 will receive 2g Oral DS107 daily. Treatment Arm 3 will receive placebo daily.

The primary objective of the study is to assess the efficacy and safety of daily 1g and 2g doses of Oral DS107 versus placebo.

Subjects will come to the clinic on 7 occasions: Screening, Baseline, Week 2, Week 4, Week 6, Week 8 (end of treatment/early termination) and Week 10 (follow-up). The primary efficacy variable will be the IGA (Investigator's Global Assessment). Secondary efficacy variables will include IGA, EASI (Eczema Area and Severity Index), and NRS (Numeric Rating Scale),

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinically confirmed diagnosis of active Atopic Dermatitis according to Hanafin and Rajka criteria
* Subjects with moderate to severe Atopic Dermatitis at baseline as defined by an IGA of minimum 3 at baseline
* Subjects with Atopic Dermatitis covering a minimum 10% of the body surface area at baseline
* Male or female subjects who are aged 18 years and older on the day of signing the informed consent form (ICF)

Exclusion Criteria:

* Subjects with other skin conditions that might interfere with Atopic Dermatitis diagnosis and/or evaluation (such as psoriasis or current active viral, bacterial and fungal skin infections) as assessed by the Investigator
* Subjects who have used systemic treatments (other than biologics) that could affect Atopic Dermatitis less than 4 weeks prior to baseline visit (Day 0), e.g. retinoids, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine and oral/injectable corticosteroids. Intranasal corticosteroids and inhaled corticosteroids for stable medical conditions are allowed
* Subjects who have used any topical medicated treatment for Atopic Dermatitis two weeks prior to start of treatment/Baseline (Day 0), including but not limited to, topical corticosteroids, tars and bleach
* Subjects who use topical products containing urea, ceramides or hyaluronic acid two weeks prior to Baseline
* Subjects who have a history of hypersensitivity to any substance in Oral DS107 or placebo capsules
* Subjects who have any clinically significant controlled or uncontrolled medical condition or laboratory abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with the interpretation of study results
* Subjects with significant uncontrolled cardiovascular, neurologic, malignant, psychiatric, respiratory or hypertensive disease, as well as diabetes and arthritis or any other illness that, in the opinion of the investigator, is likely to interfere with completion of the study
* Subjects with chronic infectious disease (e.g. hepatitis B, hepatitis C or infection with human immunodeficiency virus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weissbach, Ph.D, Study Chair — DS Biopharma
Locations (2):
- DS Biopharma Site, Philadelphia, Pennsylvania, United States
- DS Biopharma Site, Cape Town, South Africa

REFERENCES:
- [Background] Amagai Y, Oida K, Matsuda A, Jung K, Kakutani S, Tanaka T, Matsuda K, Jang H, Ahn G, Xia Y, Kawashima H, Shibata H, Matsuda H, Tanaka A. Dihomo-gamma-linolenic acid prevents the development of atopic dermatitis through prostaglandin D1 production in NC/Tnd mice. J Dermatol Sci. 2015 Jul;79(1):30-7. doi: 10.1016/j.jdermsci.2015.03.010. Epub 2015 Apr 6. PMID 25907057
- [Background] Ashcroft DM, Dimmock P, Garside R, Stein K, Williams HC. Efficacy and tolerability of topical pimecrolimus and tacrolimus in the treatment of atopic dermatitis: meta-analysis of randomised controlled trials. BMJ. 2005 Mar 5;330(7490):516. doi: 10.1136/bmj.38376.439653.D3. Epub 2005 Feb 24. PMID 15731121
- [Background] Bos JD, Kapsenberg ML, Smitt JH. Pathogenesis of atopic eczema. Lancet. 1994 May 28;343(8909):1338-41. doi: 10.1016/s0140-6736(94)92473-2. No abstract available. PMID 7910330
- [Background] Charman CR, Venn AJ, Williams HC. The patient-oriented eczema measure: development and initial validation of a new tool for measuring atopic eczema severity from the patients' perspective. Arch Dermatol. 2004 Dec;140(12):1513-9. doi: 10.1001/archderm.140.12.1513. PMID 15611432
- [Background] Desbois AP, Lawlor KC. Antibacterial activity of long-chain polyunsaturated fatty acids against Propionibacterium acnes and Staphylococcus aureus. Mar Drugs. 2013 Nov 13;11(11):4544-57. doi: 10.3390/md11114544. PMID 24232668
- [Background] Carpenter JR, Roger JH, Kenward MG. Analysis of longitudinal trials with protocol deviation: a framework for relevant, accessible assumptions, and inference via multiple imputation. J Biopharm Stat. 2013;23(6):1352-71. doi: 10.1080/10543406.2013.834911. PMID 24138436
- [Background] Williams H, Flohr C. How epidemiology has challenged 3 prevailing concepts about atopic dermatitis. J Allergy Clin Immunol. 2006 Jul;118(1):209-13. doi: 10.1016/j.jaci.2006.04.043. Epub 2006 Jun 9. PMID 16815157
- [Background] Kawashima H, Tateishi N, Shiraishi A, Teraoka N, Tanaka T, Tanaka A, Matsuda H, Kiso Y. Oral administration of dihomo-gamma-linolenic acid prevents development of atopic dermatitis in NC/Nga mice. Lipids. 2008 Jan;43(1):37-43. doi: 10.1007/s11745-007-3129-2. Epub 2007 Nov 6. PMID 17985168
- [Background] Silverberg JI, Hanifin JM. Adult eczema prevalence and associations with asthma and other health and demographic factors: a US population-based study. J Allergy Clin Immunol. 2013 Nov;132(5):1132-8. doi: 10.1016/j.jaci.2013.08.031. Epub 2013 Oct 4. PMID 24094544
- [Background] Simpson EL. Atopic dermatitis: a review of topical treatment options. Curr Med Res Opin. 2010 Mar;26(3):633-40. doi: 10.1185/03007990903512156. PMID 20070141
- [Background] Suarez AL, Feramisco JD, Koo J, Steinhoff M. Psychoneuroimmunology of psychological stress and atopic dermatitis: pathophysiologic and therapeutic updates. Acta Derm Venereol. 2012 Jan;92(1):7-15. doi: 10.2340/00015555-1188. PMID 22101513
- [Background] Kapp A. The role of eosinophils in the pathogenesis of atopic dermatitis--eosinophil granule proteins as markers of disease activity. Allergy. 1993 Jan;48(1):1-5. doi: 10.1111/j.1398-9995.1993.tb02167.x. PMID 8457021
- [Background] Leung DY, Bieber T. Atopic dermatitis. Lancet. 2003 Jan 11;361(9352):151-60. doi: 10.1016/S0140-6736(03)12193-9. PMID 12531593
- [Background] Eichenfield LF, Tom WL, Berger TG, Krol A, Paller AS, Schwarzenberger K, Bergman JN, Chamlin SL, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Margolis DJ, Silverman RA, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 2. Management and treatment of atopic dermatitis with topical therapies. J Am Acad Dermatol. 2014 Jul;71(1):116-32. doi: 10.1016/j.jaad.2014.03.023. Epub 2014 May 9. PMID 24813302
- [Background] Gutfreund K, Bienias W, Szewczyk A, Kaszuba A. Topical calcineurin inhibitors in dermatology. Part I: Properties, method and effectiveness of drug use. Postepy Dermatol Alergol. 2013 Jun;30(3):165-9. doi: 10.5114/pdia.2013.35619. Epub 2013 Jun 20. PMID 24278069
- [Background] Reynolds NJ, Franklin V, Gray JC, Diffey BL, Farr PM. Narrow-band ultraviolet B and broad-band ultraviolet A phototherapy in adult atopic eczema: a randomised controlled trial. Lancet. 2001 Jun 23;357(9273):2012-6. doi: 10.1016/S0140-6736(00)05114-X. PMID 11438134
- [Background] Iversen L, Fogh K, Kragballe K. Effect of dihomogammalinolenic acid and its 15-lipoxygenase metabolite on eicosanoid metabolism by human mononuclear leukocytes in vitro: selective inhibition of the 5-lipoxygenase pathway. Arch Dermatol Res. 1992;284(4):222-6. doi: 10.1007/BF00375798. PMID 1329675
- [Background] Kawashima H, Toyoda-Ono Y, Suwa Y, Kiso Y. Subchronic (13-week) oral toxicity study of dihomo-gamma-linolenic acid (DGLA) oil in rats. Food Chem Toxicol. 2009 Jun;47(6):1280-6. doi: 10.1016/j.fct.2009.03.001. Epub 2009 Mar 9. PMID 19275928
- [Background] Futamura M, Leshem YA, Thomas KS, Nankervis H, Williams HC, Simpson EL. A systematic review of Investigator Global Assessment (IGA) in atopic dermatitis (AD) trials: Many options, no standards. J Am Acad Dermatol. 2016 Feb;74(2):288-94. doi: 10.1016/j.jaad.2015.09.062. Epub 2015 Dec 11. PMID 26685719
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575
- [Background] Phan NQ, Blome C, Fritz F, Gerss J, Reich A, Ebata T, Augustin M, Szepietowski JC, Stander S. Assessment of pruritus intensity: prospective study on validity and reliability of the visual analogue scale, numerical rating scale and verbal rating scale in 471 patients with chronic pruritus. Acta Derm Venereol. 2012 Sep;92(5):502-7. doi: 10.2340/00015555-1246. PMID 22170091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 300 patients (100 per treatment group) with moderate to severe Atopic Dermatitis (AD) were to be included in this study.
Pre-assignment Details: Eligible patients were randomized (1:1:1) to receive 1 g DS107, 2 g DS107, or placebo administered orally once daily for 8 weeks.
Period: Overall Study
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Started | 105 | 112 | 104
Completed | 85 | 87 | 91
Not Completed | 20 | 25 | 13
Not completed — Unacceptable Adverse Events (AEs) | 0 | 3 | 1
Not completed — Patient Decision (Withdrawal of Consent to Participate) | 6 | 10 | 4
Not completed — Investigator Discretion | 0 | 2 | 1
Not completed — Lost to Follow-up | 8 | 6 | 3
Not completed — Lack of Efficacy | 5 | 3 | 3
Not completed — Other - Subject discontinued following database lock. | 1 | 0 | 0
Not completed — Other - Subject underwent knee surgery and stopped taking study medication. | 0 | 1 | 0
Not completed — Subject moved out of the country. | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consists of all patients who were randomized to the study and received at least one dose of study drug. FAS was the primary analysis population for efficacy endpoints. Analysis was done according to the actual treatment received. Demographic information used for Baseline characteristics was reported on using the Full Analysis (n=311) and Safety Analysis total was used for Participant flow (n=321).
Groups:
- Treatment Group A: 1g DS107 (2 DS107 capsules and 2 placebo capsules) orally administered once-daily for 8 weeks.
- Treatment Group B: 2g DS107 (4 DS107 capsules) orally administered once-daily for 8 weeks.
- Treatment Group C: Placebo (4 placebo capsules) orally administered once-daily for 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A | Treatment Group B | Treatment Group C | Total
Number analyzed (Participants) | 102 | 107 | 102 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (15.40) | 44.3 (16.42) | 43.3 (16.28) | 44.5 (16.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 61 | 67 | 176
  Male | 54 | 46 | 35 | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 3
  Asian | 4 | 1 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 40 | 45 | 46 | 131
  White | 52 | 55 | 46 | 153
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving an Investigators Global Assessment (IGA) of 0 (Clear) or 1 (Almost Clear) and a Decrease of at Least 2 Points in IGA in Treated Population Compared to Placebo Population at Week 8.
Description: Proportion of patients achieving an IGA of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to placebo population at Week 8. The IGA scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). IGA uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: 8 weeks
Population: The Full Analysis Set (FAS) consists of all patients who were randomized to the study and received at least one dose of study drug. FAS was the primary analysis population for efficacy endpoints. Analysis was done according to the actual treatment received.
Measure: Number; unit: Proportion of participants
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Number analyzed (Participants) | 102 | 107 | 102
Proportion of participants | 0.35 | 0.29 | 0.33
Statistical Analysis 1: Comparison: 1g DS107 vs Placebo; Test type: Superiority; p = 0.5570, General Linear Model
Statistical Analysis 2: Comparison: 2g DS107 vs Placebo; Test type: Superiority; p = 0.8774, General Linear Model

2. Secondary Outcome: Proportion of Patients Achieving an IGA Score of 0 (Clear) or 1 (Almost Clear) and a Decrease of at Least 2 Points in IGA in Treated Population Compared to Placebo Population From Baseline to Weeks 2, 4, 6, and 10.
Description: Proportion of patients achieving an IGA score of 0 (clear) or 1 (almost clear) and a decrease of at least 2 points in IGA in treated population compared to placebo population from Baseline to Weeks 2, 4, 6, and 10. The IGA scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). IGA uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: Baseline, Week 2, Week 4, Week 6 and Week 10
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Number analyzed (Participants) | 102 | 107 | 102
Proportion of participants
  Week 2 | 0.02 | 0.00 | 0.01
  Week 4 | 0.07 | 0.03 | 0.06
  Week 6 | 0.15 | 0.19 | 0.16
  Week 10 | 0.32 | 0.31 | 0.43

3. Secondary Outcome: Proportion of Patients Achieving a Decrease of at Least 2 Points in IGA in Treated Population Compared to Placebo Population From Baseline to Weeks 2, 4, 6, 8, and 10
Description: Proportion of patients achieving a decrease of at least 2 points in IGA in treated population compared to placebo population from Baseline to Weeks 2, 4, 6, 8, and 10. The IGA scale awards a score of 0-4 based on a 5-point severity scale from clear to severe disease (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease). IGA uses clinical characteristics of erythema, infiltration, papulation and oozing/crusting as scoring guidelines for the overall severity assessment.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8 and Week 10
Population: as for outcome 1
Measure: Number; unit: Proportion of participants
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Number analyzed (Participants) | 102 | 107 | 102
Proportion of participants
  Week 2 | 0.03 | 0.02 | 0.03
  Week 4 | 0.08 | 0.07 | 0.08
  Week 6 | 0.18 | 0.21 | 0.20
  Week 8 | 0.38 | 0.31 | 0.34
  Week 10 | 0.34 | 0.31 | 0.41

4. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) in Treated Population Compared to Placebo Population at Weeks 2, 4, 6, 8, and 10
Description: Change from Baseline in EASI in treated population compared to placebo population at Weeks 2, 4, 6, 8, and 10. It quantifies the severity of a patient's AD based on both lesion severity and the percent of Body Surface Area (BSA) affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately, half points are permitted) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The subscales used are summed in order to give a final EASI score. A decrease in EASI score represents a positive outcome for the patient.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8 and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: EASI Index
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Number analyzed (Participants) | 102 | 107 | 102
EASI Index
  Week 2 | -3.97 (6.932) | -2.94 (6.120) | -2.62 (4.106)
  Week 4 | -7.64 (7.366) | -6.06 (6.018) | -6.86 (6.656)
  Week 6 | -9.66 (7.913) | -8.64 (6.863) | -8.85 (8.599)
  Week 8 | -11.73 (8.894) | -9.59 (9.322) | -11.03 (8.852)
  Week 10 | -12.15 (9.205) | -10.34 (7.513) | -11.56 (8.918)

5. Secondary Outcome: Change From Baseline in Numeric Rating Scale (NRS) for Pruritus in Treated Population Compared to Placebo Population at Weeks 2, 4, 6, 8, and 10
Description: Change from Baseline in Numeric Rating Scale (NRS) for pruritus in treated population compared to placebo population at Weeks 2, 4, 6, 8, and 10. Severity of pruritus related to AD will be self-assessed by patients daily using the NRS. Patients were asked to estimate the intensity of pruritus at its worst over the previous 24 hours. The Pruritus NRS is a single-question assessment tool that will be used to assess the patient's worst itch as a result of AD in the previous 24 hours. Patients scored their pruritus due to AD on a scale of 0 - 10, with 0 (no itch) and 10 (worst itch imaginable). Patients will complete the rating scale at screening and then daily starting at baseline through to the last study visit. A decrease in NRS represents a positive outcome for the patient.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8 and Week 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1g DS107 | 2g DS107 | Placebo
Number analyzed (Participants) | 102 | 107 | 102
score on a scale
  Week 2 | -1.0 (1.74) | -1.3 (1.61) | -1.3 (1.98)
  Week 4 | -1.8 (1.97) | -2.2 (2.18) | -2.2 (2.47)
  Week 6 | -2.4 (2.15) | -2.7 (2.38) | -2.7 (2.54)
  Week 8 | -2.9 (2.41) | -3.2 (2.53) | -3.3 (2.86)
  Week 10 | -3.5 (2.56) | -3.4 (2.94) | -3.6 (2.84)

ADVERSE EVENTS:
Time Frame: 10 weeks.
Description: Any undesirable experience occurring to a patient who has received at least one dose of study drug, whether or not considered related to the Investigational Medicinal Product(s) (IMP(s)).
Arm/Group | 1g DS107 | 2g DS107 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/112 | 0/104
Serious Adverse Events (participants affected / at risk) | 1/105 | 1/112 | 0/104
Other Adverse Events (participants affected / at risk) | 34/105 | 42/112 | 34/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1g DS107 (N=105) | 2g DS107 (N=112) | Placebo (N=104)
Hip Arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1g DS107 (N=105) | 2g DS107 (N=112) | Placebo (N=104)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Eye Pain (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 6 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 2
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 4
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 2
Vessel Puncture Site Bruise (General disorders) | 0 | 1 | 0
Food Allegry (Immune system disorders) | 0 | 0 | 1
Breast Abscess (Infections and infestations) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Eczema Infected (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 1 | 3 | 0
Oral Candidiasis (Infections and infestations) | 2 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 2 | 4
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 2
Viral Rash (Infections and infestations) | 1 | 0 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Abnormal (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Abnormal (Investigations) | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0
Bacterial Test Positive (Investigations) | 0 | 1 | 0
Blood Creatine Phosphokinase (Investigations) | 1 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 1
Blood Creatinine Increased (Investigations) | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 0 | 1 | 1
Blood Uric Acid Increased (Investigations) | 0 | 1 | 0
Crystal Urine (Investigations) | 0 | 1 | 0
Protein Urine (Investigations) | 0 | 1 | 0
Urinary Sediment Present (Investigations) | 0 | 1 | 0
Urine Uric Acid (Investigations) | 0 | 0 | 1
White Blood Cells Urine Positive (Investigations) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 5 | 7
Migraine (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Breast Tenderness (Reproductive system and breast disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 | 5 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Breast Conserving Surgery (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT02864498/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/98/NCT02864498/SAP_001.pdf